CLINICAL TRIAL: NCT06720480
Title: Thalassaemia Severity Score in Upper Egypt Patients Attending Assuit University Children Hospital
Brief Title: Thalassaemia Severity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzhraa gaber mohamed, Resident doctor, Assiut University
Other Study IDs: Thalassaemia severity
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Thalassaemia
Keywords: Thalassaemia severity score
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Homglobin Electrophoresis — To diagnose thalassaemia &best method to control disease progress

SUMMARY:
This study aims to develop a nuanced understanding of thalassemia severity in Upper Egypt by integrating various clinical parameters beyond transfusion frequency. By doing so, it seeks to enhance patient management and ultimately improve quality of life for those affected by this condition.

DETAILED DESCRIPTION:
Thalassemia syndrome classified as hemoglobinopathies, represent one of the most prevalent classes of single-gene disorders globally. The mutations in the HBB gene lead to variable impacts on the production of globin proteins, which in turn affects the overall function of hemoglobin. The genetic variants contribute significantly to the diverse clinical presentations and severity of thalassemia. Traditionally, thalassemia has been categorized into Major, intermediate, and Minor based on the frequency of blood transfusions required for survival It has been observed that anemia may not be the sole determinant of thalassemic disease severity, other factors are also responsible for overall clinical status.

Accordingly, clinical conditions of the thalassemia patient, cannot classified based on the transfusion status.

Phadke et al. (2006), proposed a classification that considers multiple parameters beyond transfusion status . Similarly, Sripichai et al , (2008) classified HbE/β-thalassemia into the 3 categories of mild, moderate, and severe. Another classification was also introduced by Thalassemia International Federation (TIF) , which 'was bit modification Sripichai et al 2008 . Despite these advancements, existing classifications still tend to simplify thalassemia into three categories Globally, An estimated 1-5% of the global population are carriers of a genetic thalassemia mutation.Although the epidemiology of the various clinical forms remains poorly recognized, the disease is known to be highly prevalent in the area extending from sub-Saharan Africa, through the Mediterranean region and Middle East, to the Indian subcontinent and East and Southeast Asia.Thus, >90% of patients with these disorders live in low- and middle-income countries

ELIGIBILITY:
Inclusion Criteria:

- Children and adolescents aged from 18 month to 18 year old. Those with thalassemia

Exclusion Criteria:

* Non Thalassaemia children

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 6month till 18years who have thalassaemia
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Scoring thalassaemia severity | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Mansour Galal, Associate professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Danjou F, Francavilla M, Anni F, Satta S, Demartis FR, Perseu L, Manca M, Sollaino MC, Manunza L, Mereu E, Marceddu G, Pissard S, Joly P, Thuret I, Origa R, Borg J, Forni GL, Piga A, Lai ME, Badens C, Moi P, Galanello R. A genetic score for the prediction of beta-thalassemia severity. Haematologica. 2015 Apr;100(4):452-7. doi: 10.3324/haematol.2014.113886. Epub 2014 Dec 5. PMID 25480500